CLINICAL TRIAL: NCT04184505
Title: Prospective Randomized Study on the Feasibility of Allogeneic Stem Cell Transplantation in Higher-risk-myelodysplastic Syndromes, Performed Upfront or Preceded by Azacitidine or Conventional Chemotherapy According to the BM-blast Proportion
Brief Title: Feasibility of Allogeneic Stem Cell Transplantation in Higher-risk-MDS (ACROBAT)
Acronym: ACROBAT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDS0519
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: High-risk MDS
Keywords: MDS; Transplant; Azacitidine
MeSH Terms: interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard clinical treatment (Active Comparator): If BM-blasts >= 10%: Conventional chemotherapy: induction one cycle (3+7 protocol) and one optional consolidation cycle, followed by HSCT if a suitable sibling or unrelated donor is available versus
  If BM blasts are <10%: HSCT upfront
  Interventions: Drug: Standard Chemotherapy; Procedure: Allogeneic stem cell transplantation
- Experimental treatment (Experimental): If BM-blasts >= 10%: Azacitidine (AZA) 75mg/sqm/day subcutaneously for 7 days every 28 days (1 cycle of 28 days) for at least 4 cycles, followed by HSCT if a suitable sibling or unrelated donor is available
  If BM blasts are <10%: Azacitidine (AZA) 75mg/sqm/day subcutaneously for 7 days every 28 days (1 cycle of 28 days) for at least 4 cycles, followed by HSCT if a suitable sibling or unrelated donor is available
  Interventions: Drug: Azacitidine; Procedure: Allogeneic stem cell transplantation

INTERVENTIONS:
Drug: Azacitidine — 75mg/mq/day subcutaneously for 7 days every 28 days
  Other Names: AZA
  Arms: Experimental treatment
Drug: Standard Chemotherapy — 1. cycle (induction): i.v. 3+7 (Citarabine 200 mg/m2 iv continuous infusion (24 h) for 7 days, Daunorubicine 60 mg/mq iv day 1-3)
  2. cycle (consolidation): i.v. 3+7 (Citarabine 200 mg/m2 iv continuous infusion (24 h) for 7 days, Daunorubicine 45 mg/mq iv day 1-3)
  Other Names: STD CHT
  Arms: Standard clinical treatment
Procedure: Allogeneic stem cell transplantation — Allogeneic stem cell transplantation
  Other Names: HSCT

SUMMARY:
Open-label, randomized multicenter phase III non-inferiority study

DETAILED DESCRIPTION:
Open-label, randomized, prospective multicenter phase III study to compare the role of HMT followed by HSCT vs HSCT upfront in HR-MDS with <10% of BM blasts and of CHT vs HMT followed by HSCT in HR-MDS with >10% BM blasts in terms of feasibility of HSCT (non-inferiority trial).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed higher-risk MDS, including IPSS Intermediate-2 and high, and IPSS-R intermediate to very-high
2. Age 18-70 years
3. Previously untreated for HR-MDS
4. HSCT - eligible
5. Life expectancy ≥3 months;
6. Signed written informed consent according to ICH/EU/GCP and national local laws
7. Eastern Cooperative Oncology Group Performance Status Grade of 0-2

Exclusion Criteria:

1. Acute myeloid leukaemia with >20% blasts in BM or peripheral blood (PB);
2. concurrent malignancy diagnosed in the past 12 months (with the exception of skin basalioma);
3. severe renal, cardiac, liver or lung impairment;
4. pregnant or lactating or potentially fertile (both males and females), who have not agreed to avoid pregnancy during the trial period; Women of childbearing potential and men must agree to use effective contraception during and up to 3 months after treatment with azacitidine.
5. HIV infection; active, uncontrolled HCV or HBV infections or liver cirrhosis;
6. clinically relevant neurological or psychiatric diseases;
7. hypersensitivity (known or suspected) to AZA;
8. prior Treatments:

   1. prior investigational drugs (within 30 days);
   2. radiotherapy, chemotherapy, or cytotoxic therapy for non-MDS conditions within the previous 6 months;
   3. growth factors (EPO, G-CSF or GM-CSF) during the previous 21 days;
   4. androgenic hormones during the previous 14 days;
   5. prior transplantation or cytotoxic therapy, including azacitidine, AZA or chemotherapy, administered to treat MDS (a previous treatment with Lenalidomide is admitted, provided that lenalidomide had been stopped at least 60 days before enrolment).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of HSCT in terms of proportion of patients who receive HSCT of the total number of randomized patients | 4 years
  Split patients in two categories: the feasibility of HSCT (ITT) in patients with HR-MDS with a proportion of bone marrow blasts below 10% and in patients with a proportion of BM blasts equal or greater than 10%.

CONTACTS AND LOCATIONS:
Overall Officials: Voso, Principal Investigator — AOU POLICLINICO TOR VERGATA - ROMA - UOC TRAPIANTO CELLULE STAMINALI
Locations (46):
- Italy (46):
  - 058 - Aon Ss. Antonio E Biagio E C. Arrigo - Soc Ematologia, Alessandria
  - Aou Ospedali Riuniti "Umberto I - G.M. Lancisi - G. Salesi - Sod Clinica Ematologica, Ancona
  - Presidio Ospedaliero Av5 Osp. Gen. Prov.Le "C.G.Mazzoni" - Uoc Ematologia, Ascoli Piceno
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - Aou Di Bologna - Policlinico S. Orsola-Malpighi - Uoc Ematologia, Bologna
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - Asl Brindisi, Ospedale 'Perrino'- Uo Ematologia, Brindisi
  - U.O.C. Oncoematologia - Istituto Oncologico Veneto Irccs - Presidio Ospedaliero S. Giacomo Apostolo, Castelfranco Veneto
  - Aou Policlinico Vittorio Emanuele, Po Ospedaliero "G. Rodolico" - Uo Ematologia Con Trapianto Di Midollo Osseo, Catania
  - Aou Arcispedale Sant'Anna - Cona (Fe) - Uoc Ematologia E Fisiopatologia Della Coagulazione, Cona
  - Aso S. Croce E Carle - Sc Ematologia, Cuneo
  - Aou Ospedali Riuniti- Uoc Ematologia, Foggia
  - Asl Latina, Presidio Ospedaliero Nord - Ospedale Santa Maria Goretti - Uoc Ematologia, Latina
  - Asl Lecce, Ospedale 'V. Fazzi' - Uo Ematologia, Lecce
  - Aulss 3 Serenissima, Ospedale Dell'Angelo Uo Ematologia, Mestre
  - Asst Grande Ospedale Metropolitano Niguarda - Milano - Sc Ematologia, Milan
  - Irccs Ospedale S. Raffaele - Milano - Uo Oncoematologia, Milan
  - Aou Di Modena - Sc Ematologia, Modena
  - Ao Di Rilievo Nazionale Antonio Cardarelli - Napoli - Uoc Ematologia Con Trapianto Di Midollo, Napoli
  - Aou San Luigi Gonzaga - Orbassano - Scdu Ematologia Generale E Oncoematologia, Orbassano
  - Asl Salerno, Presidio Ospedaliero Tortora Pagani - Ematologia, Pagani
  - Aou Policlinico P. Giaccone - Uo Ematologia, Palermo
  - Asl Pescara, Presidio Ospedaliero 'Spirito Santo' - Uoc Ematologia Clinica, Pescara
  - Asl Di Piacenza, Ospedale "Guglielmo Da Saliceto" - Ematologia E Centro Trapianti, Piacenza
  - Aou Pisana - Uo Ematologia Universitaria, Pisa
  - Grande Ospedale Metropolitano "Bianchi-Melacrino-Morelli" Po E. Morelli - Reggio Calabria - Uoc Ematologia, Reggio Calabria
  - Arcispedale Santa Maria Nuova, Irccs - Sc Ematologia, Reggio Emilia
  - Ausl Della Romagna, Ospedale "Infermi" - Uo Ematologia, Rimini
  - Ao Complesso Ospedaliero San Giovanni / Addolorata - Roma - Uoc Ematologia, Roma
  - Ao San Camillo Forlanini Uoc Ematologia E Trapianto Cellule Staminali, Roma
  - Aou Policlinico Tor Vergata - Roma - Uoc Trapianto Cellule Staminali, Roma
  - Aou Sant'Andrea - Roma - Uoc Ematologia, Roma
  - Asl Roma 2, Ospedale S. Eugenio- Uoc Ematologia, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs - Roma - Area Ematologica, Roma
  - Istituti Fisioterapici Ospitalieri - Ifo - Istituto Regina Elena - Roma - Uosd Ematologia, Roma
  - Policlinico Universitario Campus Bio Medico - Roma - Uoc Ematologia E Trapianto Di Cellule Staminali, Roma
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma
  - Aou "San Giovanni Di Sio E Ruggi D'Aragona" - Uoc Ematologia E Trapianti Di Cellule Staminali Emopoietiche, Salerno
  - Aou Di Sassari - Cliniche Universitarie - Stabilimento Cliniche Di San Pietro - Uoc Ematologia, Sassari
  - Aou Senese - Uoc Ematologia E Trapianti, Siena
  - Aou Citta' Della Salute E Della Scienza - Osp. S. Giovanni Battista Molinette - Sc Ematologia 2, Torino
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia - Università Degli Studi Di Torino, Torino
  - ENTE ECCLESIASTICO CARDINALE G. PANICo - UO EMATOLOGIA, Tricase
  - Asui Di Udine - Presidio Ospedaliero "Santa Maria Della Misericordia" - Clinica Ematologica, Udine
  - Aou Integrata Di Verona, Policlinico G.B. Rossi - Uoc Ematologia, Verona
  - Asl Di Viterbo, Complesso Ospedaliero Di Belcolle - Uoc Ematologia, Viterbo